CLINICAL TRIAL: NCT05813769
Title: Dairy and Plant Amino Acid Uptake. An Explorative Study
Acronym: DaPa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DaPa
Record Dates: First submitted 2023-03-27; First posted 2023-04-14 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Amino Acid Plasma Profile
Keywords: Dairy protein; Plant protein; Postprandial plasma amino acid profiles; Essential amino acids (EAA); Total amino acids (AA)
MeSH Terms: interventions — Plant Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dairy protein 1 (Active Comparator)
  Interventions: Dietary Supplement: Dairy protein
- Dairy protein 2 (Active Comparator)
  Interventions: Dietary Supplement: Dairy protein
- Plant protein 1 (Experimental)
  Interventions: Dietary Supplement: Plant protein
- Plant protein 2 (Experimental)
  Interventions: Dietary Supplement: Plant protein
- Plant protein 2 + added AA (Experimental)
  Interventions: Dietary Supplement: Plant protein
- Plant protein 2 + Dairy protein 2 (Experimental)
  Interventions: Dietary Supplement: Dairy protein; Dietary Supplement: Plant protein

INTERVENTIONS:
Dietary Supplement: Dairy protein — During each visit, research subjects will receive the product dissolved in water, representing a 20g protein load.
  Arms: Dairy protein 1; Dairy protein 2; Plant protein 2 + Dairy protein 2
Dietary Supplement: Plant protein — During each visit, research subjects will receive the product dissolved in water, representing a 20g protein load.
  Arms: Plant protein 1; Plant protein 2; Plant protein 2 + Dairy protein 2; Plant protein 2 + added AA

SUMMARY:
To optimize the environmental sustainability, a protein transition to more plant-based protein sources is required. However, the protein quality of plant-based sources is lower than that of the dairy proteins casein and whey, which contain high levels of essential amino acids. The amino acid absorption characteristics of many plant-based proteins are unknown.

The present study aims to estimate differences in postprandial plasma total essential amino acids (TEAA) profiles after protein consumption of different protein sources in blood of healthy participants. This explorative study has a randomized, cross-over, double-blind, controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women;
* Age ≥18 and ≤40 years;
* Body mass index (BMI) ≥18.5 and ≤30 kg/m2 ;
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor).

Exclusion Criteria:

* Any self-reported metabolic, gastrointestinal, inflammatory or chronic disease (such as anemia, diabetes, hepatitis, cardiovascular disease);
* Having a history of medical or surgical events that may significantly affect the study outcome;
* Anaemia (Haemoglobin (Hb) values <7.5 mmol/L for women and <8.5 mmol/L for men), as assessed by finger prick blood during screening visit;
* Having a food or protein allergy
* Use of glucose lowering drugs, insulin;
* Use of medication that may impact gastric emptying (e.g. gastric acid inhibitors or laxatives);
* Use of antibiotic treatment less than 1 month before start of the study and during the study;
* Use of anti-depressives as a treatment for depression;
* Use of protein supplements (must be stopped 1 week before the first test day);
* Reported weight loss or weight gain of > 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period;
* Reporting to follow or having planned a slimming or medically prescribed diet.
* Not willing to keep a stable lifestyle during the study period;
* Recent blood donation (<1 month prior to test day 1 of the study) or not willing to stop donation during and 1 month after the study;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Postprandial blood TEAA profiles | Frome baseline up to 5 hours postprandial
  Postprandial plasma total essential amino acids (TEAA) profiles after protein consumption, determined by appearance in blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen Food & Biobased Research, Food, Health & Consumer Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided